CLINICAL TRIAL: NCT01801228
Title: Swedish, Multicentered, Randomized Study of Eplerenone Versus Spironolactone as Treatment of Ascites Due to Liver Cirrhosis Regarding Efficacy and Side Effects
Brief Title: Eplerenone Versus Spironolactone as Treatment of Ascites Due to Liver Cirrhosis; a Study of Efficacy and Side Effects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties to include patients
Sponsor: Emma Nilsson (Other)
Collaborators: Göteborg University (Other); Uppsala University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); University Hospital, Umeå (Other); Region Örebro County (Other)
Responsible Party: Sponsor-Investigator, Emma Nilsson, Gastroenterologist, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001264-22; 2011-001264-22 (EudraCT Number)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Ascites; Cirrhosis
MeSH Terms: conditions — Ascites; Fibrosis | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Experimental): oral daily treatment with doses 100 to 400 mg
  Interventions: Drug: Eplerenone
- Spironolactone (Active Comparator): oral daily treatment with doses 100 to 400 mg
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
This study compares Spironolactone, a non-selective aldosterone antagonist, with Eplerenone, a selective aldosterone antagonist, regarding efficacy and hormonal side effects when treating male cirrhotic patients with uncomplicated ascites over a 6 month period. The investigators hypothesis is that Eplerenone is as effective as Spironolactone as treatment of ascites with less side effects such as painful gynecomastia.

ELIGIBILITY:
Inclusion Criteria:

Male Ascites Cirrhosis

-

Exclusion Criteria:

Prior treatment with aldosterone antagonist Uncontrolled heart disease or diabetes Current malignancy Current medication interacting with aldosterone antagonists

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Ascites | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Skane, Lund, Skåne County, Sweden